CLINICAL TRIAL: NCT02685592
Title: Photodynamic Therapy for Melanoma Precursor Lesion Lentigo Maligna Using 5-aminolevulinic Acid Nanoemulsion (BF-200 ALA) as a Light Sensitizing Cream
Brief Title: Photodynamic Therapy for Lentigo Maligna Using 5-aminolevulinic Acid Nanoemulsion as a Light Sensitizing Cream
Acronym: LM PDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Huslab, Finland (Unknown); Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q291dnro62/2015
Record Dates: First submitted 2016-02-13; First posted 2016-02-19 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Lentigo Maligna
Keywords: Lentigo Maligna; Photodynamic Therapy; Hyperspectral Imaging
MeSH Terms: conditions — Hutchinson's Melanotic Freckle | interventions — BF-200 ALA; Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lentigo maligna patients (Experimental): All the participants with histologically confirmed lentigo maligna will receive photodynamic therapy three times with 2 weeks' intervals. The borderline of treatment area is delineated with Wood's lamp and hyperspectral imaging system using 5 millimeter margins. Before applying the 5-aminolevulinic acid nanoemulsion (BF-200 ALA, Ameluz®) light sensitizing gel the skin of treatment area is prepared with fractional ablative CO2-laser to enhance absorption. Ameluz® is spread as a 1 millimeter thick layer on the skin. After light sensitizer absorption the treatment area is illuminated with artificial red light (Aktilite CL128 lamp) using a light dose of 90 J/cm2. Finally 4 weeks after the last PDT treatment LM is excised surgically using 5 mm margins.
  Interventions: Drug: 5-aminolevulinic acid nanoemulsion

INTERVENTIONS:
Drug: 5-aminolevulinic acid nanoemulsion — A 1 millimeter thick layer of 5-aminolevulinic acid nanoemulsion light sensitizing gel is applied on the skin and let to absorb 3 hours before illumination.
  Other Names: BF-200 ALA; Ameluz®

SUMMARY:
This study investigates the efficacy of photodynamic therapy (PDT) in the treatment of lentigo maligna (LM). Hyperspectral imaging system (HIS) will be used to determine the margins of LM and to rule out possible invasion. Participants will receive photodynamic therapy three times consecutively with intervals of two weeks using 5-aminolevulinic acid nanoemulsion (BF-200 ALA, Ameluz®) as a light sensitizing cream. Four weeks after last photodynamic therapy the lentigo maligna lesion will be excised surgically from the skin. Result of the treatment is assessed with histopathological examination and immunohistochemical staining of removed tissue specimen.

DETAILED DESCRIPTION:
Lentigo maligna (LM) is an in-situ form of melanoma which occurs on sun-exposed skin. Untreated LM can progress into invasive lentigo maligna melanoma (LMM). The incidence of LM/LMM is constantly increasing as the population grows older and lifelong sun-exposure is on the rise. Clinically it is difficult both to determine the borderline of LM as well as to differentiate LMM from LM. A novel imaging method hyperspectral imaging system (HIS) can be used for delineating margins of LM and for spotting invasion inside LM lesion. The gold standard treatment for LM is surgical excision with adequate (≥5 mm) margins. Due to large size of LM lesions and typical location on face or neck the surgical treatment is challenging and can cause aesthetic and functional deficit for the patient. Furthermore, LM patients tend to be elderly who may have anesthetic contraindications. Other treatment modalities for LM have been studied but none of them still has proved to be efficient enough. Recently, photodynamic treatment (PDT) has been suggested as a promising novel treatment method for LM.

In this prospective pilot study we investigate whether the photodynamic therapy (PDT) is effective for treatment of lentigo maligna. 10-15 patients with a histologically confirmed lentigo maligna are included in the trial. The study course is as follows: During the first visit in the clinic, the suspected LM lesion is examined clinically under Wood's lamp and imaged with a HIS camera. Elicited margins from both methods are marked on a transparent sheet and the treatment area is photographed. A biopsy is taken from the darkest-colored part of LM to confirm diagnosis and to rule out invasion. Next, the patients receive PDT treatment three times with 2 weeks' intervals. Before applying the Ameluz® light sensitizer gel the skin of treatment area is prepared with fractional ablative CO2-laser to enhance absorption. After light sensitizer absorption the LM lesion is illuminated with artificial red light (Aktilite CL128 lamp) using a light dose of 90 J/cm2. Finally 4 weeks after the last PDT treatment LM is excised surgically using 5 mm margins. The efficacy of PDT is assessed after surgical excision with histopathological examination and immunohistochemical staining (MART, Mel-5 and MITF stains). The final result of the treatment is controlled 6 months after the surgical excision.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-invasive lentigo maligna located in the skin of face, neck or upper body region

Exclusion Criteria:

* Biopsy shows invasive melanoma inside lentigo maligna lesion prior treatment
* Porphyria or solar dermatitis
* Allergy for photosensitizer (5-aminolaevulinic acid) used in study
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The histopathological and immunohistochemical curing of lentigo maligna | 2 months
  The efficacy of PDT treatment is assessed after surgical excision with histopathologic examination and immunohistochemical staining (MART, Mel-5 and MITF stains). The final result of the treatment is controlled 6 months after the surgical excision.

SECONDARY OUTCOMES:
The changes in hyperspectral images induced by photodynamic therapy | 2 months
  The lentigo maligna will be imaged with hyperspectral imaging system before and after PDT treatment. The difference in hyperspectral images will be assessed.
The occurrence of TERT-mutations in Lentigo maligna | 2 months
  The participants' will be asked a separate permission to partake in a TERT (telomerase reverse transcriptase) gene study. If permission is granted a partial tissue specimen of excised lentigo maligna lesion will be sent to Heidelberg, Germany for analysis of TERT (telomerase reverse transcriptase) gene mutations.

OTHER OUTCOMES:
The experienced pain of participants during photodynamic therapy | 1 day
  Participants will be asked to fill visual analogue scales (VAS) of pain experienced during illumination phase of photodynamic therapy.
Delayed skin reactions after photodynamic therapy | 2 days, 2 weeks
  The participants will have a nurse's appointment two days after the first PDT treatment to photograph and to evaluate the degree of delayed inflammatory skin reactions due to treatment. The skin reactions are also evaluated by the dermatologist during second and third PDT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janne Räsänen, Lic. Med., Principal Investigator — Päijät Häme Central Hospital; Mari Grönroos, D. Med. Sc., Study Director — Päijät Häme Central Hospital; Noora Neittaanmäki-Perttu, D. Med. Sc., Study Chair — HUSLAB; Mari Salmivuori, Lic. Med., Study Chair — Päijät Häme Central Hospital; Leila Jeskanen, Lic. Med., Study Chair — HUSLAB; Erna Snellman, Professor, Study Chair — Tampere University
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Finland

IPD SHARING:
Plan to Share IPD: No